CLINICAL TRIAL: NCT02959528
Title: The Effects of Working Memory Training in Children With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, I-hsuan Shen, Associated professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-5308A3
Record Dates: First submitted 2016-10-31; First posted 2016-11-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Psychophysiology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): ADHD group treated with visual-perceptual training
  Interventions: Other: perceptual training
- Experiment (Experimental): ADHD group treated with working memory training
  Interventions: Other: Working memory training

INTERVENTIONS:
Other: Working memory training — n-back training program
  Arms: Experiment
Other: perceptual training — visual-perceptual training program
  Arms: Control

SUMMARY:
Previous studies indicated that children with attention-deficit/hyperactivity disorder (ADHD) often suffer from deficits in executive function, such as attentional control, inhibition, and working memory. One of these executive functions, working memory, plays a critical role in academic performance and classroom behavior. Working memory is essential for performing complex cognitive tasks such as comprehension, learning, and reasoning. Several studies have shown that training of working memory has positive effects for ADHD and other cognitive disorder in children. However, transfer effects across studies appear to be variable and inconsistent. Event-related potentials can be a useful tool to gain insights into such mechanism. Therefore, the aim of the present study is to investigate both near and far transfer effects of N-back training in children with ADHD. In addition, the recording and analysis of event-related potentials will be adopted while children with ADHD perform the complex visuo-spatial and phonological working memory tasks.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosed according to criteria specified in Diagnostic and statistical manual of mental disorders (DSM-5)
* aged between 8 and 10 years
* intelligence quotient > 80 (based on Test of Nonverbal Intelligence-Third Edition)
* had normal or corrected-to-normal vision
* right-handed

Exclusion Criteria:

* diagnosis of clinically significant oppositional defiant disorder, Autistic Spectrum Disorders, Asperger's syndrome or depression
* history of seizures

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11-25 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Automated Working Memory Assessment | 6 weeks
  Visuospatial working memory change after intervention measured by Automated Working Memory Assessment

SECONDARY OUTCOMES:
Working memory index in Wechsler Intelligence Scale for Children-IV | 6 weeks
  Verbal working memory change after intervention measured by Working memory index in WISC-IV
Event-related potentials | 6 weeks
  Event-related potentials are measured brain response on effects of working memory training

CONTACTS AND LOCATIONS:
Overall Officials: I-Hsuan Shen, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No